CLINICAL TRIAL: NCT05793541
Title: Micro-randomized Trial to Assess Brief, Just-in-time Interventions for Reducing Short-term Suicide Risk
Brief Title: Just-in-time Interventions for Reducing Short-term Suicide Risk
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: University of Michigan (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Rebecca G. Fortgang, Ph.D., Assistant Professor, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023P000595
Record Dates: First submitted 2023-03-20; First posted 2023-03-31 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Suicide
Keywords: Suicide; Suicidal Thoughts; Micro-Randomized Trial; Ecological Momentary Assessment; Just-in-Time Intervention
MeSH Terms: conditions — Suicide; Suicidal Ideation

STUDY DESIGN:
Intervention Model Description: During the four weeks following discharge from psychiatric hospitalization for suicidal thoughts or behaviors, participants will be prompted to complete up to 4 brief smartphone surveys per day that assess current suicidal urges and intent on a 0 to 10 scale. After each completed survey, participants will be "micro-randomized" to one of several brief just-in-time interventions. Both the intervention method (phone call from a clinician, text messaging from a clinician, automated interactive smartphone-based tool, or automated non-interactive pop-up messages) and intervention content (reminder to either use their safety plan [any and all included components] or a specific component of their safety plan) will be randomized according to the current level of suicidal urges and intent.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Just-in-time intervention for promoting use of the safety plan or its components (Experimental): Completed surveys will be assigned to a risk level (High Risk, Medium/Low Risk, or No Risk) based on self-reported level of suicidal urge and intent. Participants will be "micro-randomized" to one of the available intervention options based on the survey's risk level. All interventions will include reminders to use the safety plan or its components. At High Risk, participants will be randomized to either receive a phone call from a clinician, text messaging from a clinician, or automated interactive smartphone tool. At Medium/Low risk, participants will be randomized to receive an automated interactive smartphone tool, non-interactive pop-up messages, or no intervention. No randomization will occur (and no intervention given) at No Risk.
  Interventions: Behavioral: Phone call; Behavioral: Text messaging; Behavioral: Automated interactive smartphone-based tool; Behavioral: Non-interactive pop-up messages

INTERVENTIONS:
Behavioral: Phone call — A phone call from a trained study clinician that uses a standardized phone script to (a) conduct a risk assessment and (b) recommend that the participant use their safety plan (any and all included components), which will be reviewed and revised as-needed during the call. This intervention occurs at High Risk only.
Behavioral: Text messaging — A text message conversation initiated by a trained study clinician that uses a standardized text messaging script to (a) conduct a risk assessment and (b) recommend that the participant use their safety plan (any and all included components), which will be reviewed and revised as-needed during the text messaging interaction. This intervention occurs at High Risk only.
Behavioral: Automated interactive smartphone-based tool — An automated interactive, smartphone-based tool that will (a) (at High Risk only) guide the participant through a risk assessment and (b) (at High and Medium/Low Risk) present recommendation to use and a review of the safety plan.
Behavioral: Non-interactive pop-up messages — Automated non-interactive, static pop-up messages that recommend use of the safety plan or its components (Medium/Low Risk only).

SUMMARY:
The goal of this study is to test the effects of just-in-time intervention strategies aimed to promote implementation of the safety plan and its components at different levels of suicidal urges and intent. The main questions the investigators aim to answer are:

1. What is the acceptability and feasibility of the just-in-time intervention strategies?
2. What are the proximal effects of just-in-time intervention strategies aimed to promote use of the safety plan and its components?
3. What internal and external contextual factors moderate the just-in-time intervention effects?

Participants (adults hospitalized for suicidal thoughts or behaviors) will:

* Answer questions about current suicidal thoughts on their smartphone up to 4 times each day during both hospitalization and the 4 weeks after they leave the hospital
* Each time they submit a survey, be immediately randomized to receive (or not receive) a just-in-time intervention tailored to their level of current suicidal thoughts
* Answer brief follow-up questions on their smartphone within a couple hours of each randomization
* Provide feedback on their experience with the just-in-time interventions

DETAILED DESCRIPTION:
As the 12th leading cause of death in the United States, suicide is an alarmingly prevalent public health problem. The time period of highest risk for suicide and related behavior (SRB) is immediately (e.g., the weeks) following psychiatric hospitalization. Effective and scalable strategies for preventing SRB among individuals recently discharged from inpatient treatment are urgently needed. Encouragingly, brief evidence-based interventions now exist that reduce risk for suicide after acute psychiatric care. A primary example is safety planning, which involves developing a prioritized list of coping strategies and sources of support that people can use to mitigate future suicidal crises; this intervention is now recommended as part of standard inpatient clinical care. However, it has been shown that well over one-third of suicidal patients who have a safety plan never use it. Additionally, little is known about when (and for whom) specific components of the safety plan, which includes internal coping strategies, social support activities, and help-seeking behaviors, are most accessible and effective. Optimizing real-world safety plan use with scalable intervention strategies delivered via mobile technology has great potential to improve the effectiveness of an already promising intervention and advance precision treatment for high-risk individuals.

This project will employ the recently developed micro-randomized trial (MRT) design to test the effectiveness of brief, just-in-time interventions aimed to promote real-world use of the safety plan and its specific components. Both the method (e.g., phone call or text messaging by a human or automated forms of smartphone-based messaging) and content (e.g., recommendation to use the safety plan in its entirety or a specific component) will be randomized according to individuals' current levels of suicidal urges and intent. Participants will be psychiatric inpatients admitted for suicidal thoughts or behaviors who agree to participate in an intensive longitudinal monitoring protocol involving real-time smartphone-based surveys for the 28 days after hospitalization; after each completed survey, participants will be repeatedly "micro-randomized" to one of several just-in-time interventions. The investigators will test the hypotheses that the brief just-in-time interventions will be both acceptable and feasible, and associated with increased use of safety plan components (target mechanism) and reductions in suicidal thoughts (proximal outcome) at varying levels of suicidal thoughts, and that intervention effects will vary by both intervention method and content. The investigators will also explore internal and external contextual moderators (e.g., affect, social support) of proximal intervention effects, and collect qualitative data that will inform intervention refinement as well as the future development and implementation of just-in-time adaptive interventions.

The investigators will first conduct a small pilot MRT (N=10 participants), after which qualitative feedback collected on the intervention methods, content, amount of support, timing, and triggering, as well as overall data on acceptability and feasibility, will be used to refine the interventions before the full MRT (per Question #1 outlined above). The full MRT of the refined just-in-time interventions will be conducted in N=175 participants (and answer Questions #2 and #3 above).

ELIGIBILITY:
Inclusion Criteria:

* Experiencing suicidal thoughts as part of their inpatient admission
* Access to a smartphone following discharge
* Ability to speak and write English fluently

Exclusion Criteria:

* Any factor that impairs the ability to effectively participate in the study (e.g., significant cognitive impairment, intellectual disability, presence of violent behavior, psychotic illness/symptoms determined by the treating clinician to impair ability to understand the study or provide informed consent)
* Failure to correctly answer all true/false questions in the consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Estimated)
Dates: Start 2024-11-19 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Self-reported safety plan and coping strategy use | Within two hours of each micro-randomization
  Participants will be prompted within two hours of each micro-randomization to complete a brief follow-up smartphone survey that assesses safety plan and/or coping strategy use since the initial survey prompting micro-randomization.
Self-reported momentary suicidal urges and intent | Within two hours of each micro-randomization
  Participants will be prompted within two hours of each micro-randomization to complete a brief follow-up smartphone survey that assesses momentary suicidal urge and intent (on a 0 to 10 scale).

SECONDARY OUTCOMES:
Objective indicator of safety plan viewing | Within two hours of each micro-randomization
  The app used for real-time assessments and to deploy the just-in-time interventions will also capture whether or not the participant opened their safety plan.

OTHER OUTCOMES:
Suicide attempt | 28 days after hospital discharge
  The distal outcome of whether or not a suicide attempt occurs during the 28 days after hospital discharge will be captured via nightly smartphone-based self-report survey and manual review of electronic health records.
Hospital visit for suicidal thoughts or suicide-related behavior (SRB) | 28 days after hospital discharge
  The distal outcome of whether or not a hospital visit occurs for suicidal thoughts or SRB during the 28 days after hospital discharge will be captured via nightly smartphone-based self-report survey and manual review of electronic health records.

CONTACTS AND LOCATIONS:
Locations (1):
- Mass General Brigham, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Chung DT, Ryan CJ, Hadzi-Pavlovic D, Singh SP, Stanton C, Large MM. Suicide Rates After Discharge From Psychiatric Facilities: A Systematic Review and Meta-analysis. JAMA Psychiatry. 2017 Jul 1;74(7):694-702. doi: 10.1001/jamapsychiatry.2017.1044. PMID 28564699
- [Background] Chung D, Hadzi-Pavlovic D, Wang M, Swaraj S, Olfson M, Large M. Meta-analysis of suicide rates in the first week and the first month after psychiatric hospitalisation. BMJ Open. 2019 Mar 23;9(3):e023883. doi: 10.1136/bmjopen-2018-023883. PMID 30904843
- [Background] Doupnik SK, Rudd B, Schmutte T, Worsley D, Bowden CF, McCarthy E, Eggan E, Bridge JA, Marcus SC. Association of Suicide Prevention Interventions With Subsequent Suicide Attempts, Linkage to Follow-up Care, and Depression Symptoms for Acute Care Settings: A Systematic Review and Meta-analysis. JAMA Psychiatry. 2020 Oct 1;77(10):1021-1030. doi: 10.1001/jamapsychiatry.2020.1586. PMID 32584936
- [Background] Hedegaard H, Curtin SC, Warner M. Suicide Mortality in the United States, 1999-2019. NCHS Data Brief. 2021 Feb;(398):1-8. PMID 33663651
- [Background] Klasnja P, Hekler EB, Shiffman S, Boruvka A, Almirall D, Tewari A, Murphy SA. Microrandomized trials: An experimental design for developing just-in-time adaptive interventions. Health Psychol. 2015 Dec;34S(0):1220-8. doi: 10.1037/hea0000305. PMID 26651463
- [Background] National Action Alliance for Suicide Prevention: Transforming Health Systems Initiative Work Group. Recommended standard care for people with suicide risk: Making health care suicide safe. Washington, DC: Education Development Center, Inc.; 2018.
- [Background] Stanley B, Brown GK. Safety planning intervention: A brief intervention to mitigate suicide risk. Cognitive and Behavioral Practice. 2012; 19(2): 256-264.
- [Background] Stanley B, Chaudhury SR, Chesin M, Pontoski K, Bush AM, Knox KL, Brown GK. An Emergency Department Intervention and Follow-Up to Reduce Suicide Risk in the VA: Acceptability and Effectiveness. Psychiatr Serv. 2016 Jun 1;67(6):680-3. doi: 10.1176/appi.ps.201500082. Epub 2016 Feb 1. PMID 26828397